CLINICAL TRIAL: NCT00530101
Title: The Magnetic Resonance Imaging Evaluation of Doxorubicin Cardiotoxicity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Dr. Joel Fishman, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1177-04-806; 20043031 and 20050866
Record Dates: First submitted 2007-09-14; First posted 2007-09-17 (Estimated); Last update posted 2008-06-04 (Estimated); Status verified 2008-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Doxorubicin — This pilot study will select patients who are at increased likelihood to develop cardiotoxicity, due to borderline cardiac function at baseline, advanced age, or the anticipation of a high cumulative dose of administered doxorubicin. Patients who will receive radiation therapy to the left chest during chemotherapy (i.e., left breast cancer) will be excluded so as to eliminate possible cardiotoxic effects from radiation. CMR studies will be performed at no charge to the patient, supported by the sponsor of this study. CMR imaging will be subject to IRB approval, informed consent, and HIPAA regulations. Contrast-enhanced CMR will be obtained at three time points:
  Patients will not undergo contrast-enhanced MR unless calculated GFR is equal to or greater than 60 mL/min/1.73 m2
  Other Names: 1177-04-806

SUMMARY:
The purpose of this research study is to evaluate MR imaging in subjects receiving doxorubicin chemotherapy to see if MR can detect heart damage as well as or better than MUGA scans.

This research study is expected to enroll approximately 10 subjects over 12 months at the University of Miami / Miller School of Medicine.

DETAILED DESCRIPTION:
Doxorubicin (Adriamycin) is one of the most widely used chemotherapy agents, despite its well-known causation of cardiac toxicity. Doxorubicin causes apoptotic cell death, as shown with uptake of antimyosin antibodies on nuclear medicine studies (1,2). Myocyte damage is dose-related, and produces left ventricular dysfunction that may lead to clinically significant heart failure, especially in patients with limited cardiac reserve. An estimated 7% of patients develop doxorubicin-related congestive heart failure (CHF) after a cumulative dose of 550 mg/m2 (3).

Methods to detect and prevent doxorubicin-induced cardiotoxicity have been investigated for years. Serial evaluation of left ventricular function using Multigated Acquisition (MUGA) scans (radionuclide angiocardiography) was proposed over 20 years ago as one method for detecting cardiotoxicity (4). More sophisticated nuclear imaging (PET) has not been able to demonstrate early changes of cardiotoxicity (5). There are a number of potential indicators of early cardiotoxicity such as toxic effects on the right ventricle and on left ventricular diastolic (vs. systolic) function that MUGA is not optimally suited to demonstrate. Even earlier, an imaging manifestation of cell death could provide the first clue to impending cardiotoxicity (1,2,6). Cardiac MR (CMR) has the potential to address all of these facets of doxorubicin toxicity. Biventricular function can be assessed from cine images, and CMR is well-established as a highly reliable method for cardiac functional assessment. Of even greater potential interest, cell injury and death can be demonstrated using gadolinium enhancement, both for myocardial infarction (focal enhancement) as well as myocarditis (both focal and diffuse enhancement) (7,8). Doxorubicin toxicity may in fact share pathophysiological characteristics with myocarditis (9). It is our hypothesis that CMR will be able to show both functional and cellular (infarct, microinfarct, or myocarditis-type) effects of doxorubicin toxicity as determined during and at the conclusion of doxorubicin therapy. Specifically, we hypothesize that myocardial tissue will demonstrate a greater increase in signal (decrease in T1 after contrast administration) after chemotherapy as compared to before chemotherapy.

Methods 1. Patient Selection: Ten patients selected to receive doxorubicin for breast cancer treatment will be recruited from Oncology Services at the Sylvester Cancer Center and Jackson Memorial Hospital. This pilot study will select patients who are at increased likelihood to develop cardiotoxicity, due to borderline cardiac function at baseline, advanced age, or the anticipation of a high cumulative dose of administered doxorubicin. Patients who will receive radiation therapy to the left chest during chemotherapy (i.e., left breast cancer) will be excluded so as to eliminate possible cardiotoxic effects from radiation. CMR studies will be performed at no charge to the patient, supported by the sponsor of this study. CMR imaging will be subject to IRB approval, informed consent, and HIPAA regulations. Contrast-enhanced CMR will be obtained at three time points:

1. Prior to the first dose of doxorubicin (image characteristics will serve as control values to indicate later changes).
2. After first cycle of doxorubicin.
3. At conclusion of therapy, typically 4-6 cycles; cumulative dose of 360 to 600 mg/m2 doxorubicin.

In addition to standard screening for contraindications to MR imaging, patients will be evaluated for estimated Glomerular Filtration Rate (GFR) within 30 days prior to each MR scan. This is to avoid the rare but potential complication of Nephrogenic Systemic Fibrosis in patients with severe or end-stage renal failure who receive gadolinium MR contrast (10). GFR will be calculated from serum creatinine, patient age, gender, and race, using the MDRD GFR Calculator ( Stephen Z. Fadem, M.D.) at:

http://www.kidney.org/professionals/kdoqi/gfr_calculator.cfm

Patients will not undergo contrast-enhanced MR unless calculated GFR is equal to or greater than 60 mL/min/1.73 m2

2. Imaging: CMR will be performed on the Siemens 1.5T Sonata located at the University of Miami Outpatient Diagnostic Imaging Center. It is anticipated that each scan will require approximately 60 minutes. Three imaging planes (short axis [SA] series through the ventricles, and individual 4 chamber [4CV] and 2 chamber [2CV] views) will be utilized. Sequences will consist of:

A. Precontrast imaging:

1. T1-weighted (SA series)
2. TI scout (single mid-ventricular SA) [The TI scout sequence obtains images at multiple inversion (TI) times at a single slice level]
3. TrueFISP cine gradient echo imaging (SA series, 2CV, 4CV)

B. Postcontrast imaging: after 0.1 mmol/kg OptiMARK intravenous

1. 1 minute post-injection: TI scout (single mid-ventricular SA)
2. 2-4 minutes post-injection: Turboflash inversion recovery (single mid-ventricular SA) at serial TI values to determine time of myocardial nulling
3. 5 minutes post-injection: TI scout (single mid-ventricular SA)
4. 6-9 minutes post-injection: Turboflash inversion recovery (single mid-ventricular SA) at serial TI values to determine time of myocardial nulling
5. 10-14 minutes post-injection: Segmented IR delayed imaging using TI of myocardial signal nulling (SA series, 2CV, 4CV)
6. 15 minutes post-injection: TI scout (single mid-ventricular SA)
7. 16-19 minutes post-injection : Turboflash inversion recovery (single mid-ventricular SA) at serial TI values to determine time of myocardial nulling
8. 20 minutes post-injection: TI scout (single mid-ventricular SA)
9. 21 minutes post-injection : T1-weighted (SA series)

3. Analysis: ANOVA will be used to assess for differences in measured values of the discrete variables listed in A, B, C, and D below. Data will be analyzed for all three imaging sessions together using ANOVA, and for each pair of sessions (pretreatment vs. first cycle of doxorubicin, first cycle of doxorubicin vs. maximum cumulative dose, and pretreatment vs. maximum cumulative dose) using the paired t-test (or Wilcoxon signed-rank test if variances unequal). The MR image sets will be analyzed in random order.

A. TrueFISP cine: analysis will utilize the ARGUS software package on the Siemens system. End-diastolic and end-systolic endocardial contours will be generated using a semi-automated technique whereby initial manual contouring is followed by automated contour generation, which are then manually edited before final calculations are performed.

1. Ejection fraction (biventricular) and ventricular volumes (end-systole and end-diastole).
2. Diastolic left ventricular function I. 1/3 peak filling rate (PFR) II. 1/3 filling fraction (1/3 FF)
3. Wall motion: The AHA 17-segment model will be utilized (6 segments each at basal, mid-ventricular, and near-apical levels, and a single apical segment). A five-point scale will be assigned to each segment (normal, mildly hypokinetic, severely hypokinetic, akinetic, dyskinetic). Summed values will yield a single measure of contractility for each imaging study.

B. T1-weighted

Region-of-interest signal intensity in the myocardium will be measured in the mid-left ventricular free wall, the mid-interventricular septum, and skeletal muscle for both precontrast and postcontrast T1-weighted imaging. We will calculate a variable representing "percent enhancement" for each location as follows:

% enhancement = signal intensity (postcontrast) - signal intensity (precontrast) signal intensity (precontrast)

C. The TI scout image sets will provide a single TI value of optimal myocardial nulling as well as an exponential curve to reflect the T1 recovery of myocardium at each time point of acquisition (precontrast, 1 minute postcontrast, 5 minutes postcontrast, 15 minutes postcontrast, 20 minutes postcontrast). The TI scout will be performed at multiple time points due to the dynamic nature of tissue enhancement after gadolinium administration.

D. The turboflash inversion recovery image (mid-ventricular) will provide an alternative single TI value of optimal myocardial nulling at each time point of acquisition (2-4 minutes, 6-9 minutes, and 16-19 minutes postinjection). The turboflash inversion recovery image will be performed at multiple time points due to the dynamic nature of tissue enhancement after gadolinium administration.

E. Segmented IR delayed imaging will provide images of the entire myocardium which will be evaluated for focal myocardial signal hyperintensities, whether due to infarction or myocarditis. The optimum TI value determined from (D) above will be used. If identified, lesions will be manually contoured with use of the irregular region of interest tool on the console. The infarct size will then be calculated as total infarct area multiplied by the section thickness and the specific gravity (assumed to be 1.05 g/mL) of the myocardium.

Medical records will provide data regarding cardiac morbidity or mortality.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have breast cancer and undergoing radiation treatment with a likelihood of developing cardiotoxicity.

Exclusion Criteria:

* Healthy subjects
* Males
* Subjects under the age of 18

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2004-07; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
The purpose of this research study is to evaluate MR imaging in subjects receiving doxorubicin chemotherapy to see if MR can detect heart damage as well as or better than MUGA scans. | Over a period of 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Joel Fishman, MD, Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - University of Miami Dept of Hematology/Oncology, Miami, Florida
  - University of Miami Dept of Radiology, Miami, Florida